CLINICAL TRIAL: NCT01166841
Title: The Effect of Percutaneous Superior Venae Cava Cannulation Clamping on Cerebral Near Infrared Spectroscopy During Minimally Invasive Mitral Valve Surgery
Brief Title: The Effect of Percutaneous Superior Venae Cava Cannulation Clamping on Cerebral Near Infrared Spectroscopy in MICS
Acronym: NIRSinMICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Daniel Bainbridge, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R-10-181; 16992 (Other: REB)
Record Dates: First submitted 2010-06-08; First posted 2010-07-21 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Mitral Regurgitation
Keywords: minimally invasive cardiac surgery; cardiac surgery; near infrared spectroscopy; mitral valve repair; mitral valve replacement
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- PSVC line clamped (Experimental): Clamping of the percutaneously placed superior vena cava line placed for minimally invasive mitral valve repair/replacement.
  Interventions: Procedure: PSVC line clamped
- Unclamped PSVC (No Intervention): Unclamped percutaneously placed superior vena cava line placed for minimally invasive mitral valve repair/replacement.

INTERVENTIONS:
Procedure: PSVC line clamped — A line clamp will be placed on the PSVC line while on cardiopulmonary bypass.
  Arms: PSVC line clamped

SUMMARY:
The use of minimally invasive cardiac surgery has progressed over the last 5-10 years to allow access to the heart through a small incision in the right chest. This avoids the use of a sternotomy incision through the bone in the front of the chest. The benefits of such an approach are cosmetic (smaller incision not easily visible) and faster recovery. The minimally invasive approach also eliminates the risk of sternal wound infection. Minimally invasive cardiac surgery however poses additional challenges; one of the biggest is access to the large blood vessels which need to be cannulated to allow the heart lung machine to function. In conventional surgery, these vessels are easily accessed as they are entering or leaving the heart. In minimally invasive surgery, the cannula are placed into easily accessible arteries and veins, traditionally the femoral vessels. These vessels are smaller than those by the heart and so require smaller cannula, which provide challenges to the heart lung machine. One way around this is to use more cannulae and so cannulation of a vein in the neck is also performed. This cannula however, has been associated with neck hematoma, tearing of the vein and blood loss. While placement of the cannula in the neck is routine at LHSC now, when this surgery was first performed here 10 years ago, it was done so without the neck cannula and with no injury to patients. The purpose of this study therefore, is to more rigorously study the effect of the neck cannula on heart lung bypass, and more specifically to see if oxygen delivery to the organs, and the brain in particular is sufficient to avoid hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* Elective mitral valve repair or replacement.
* Scheduled to have minimally invasive approach (right thoracotomy)
* No contraindication to SVC line placement

Exclusion Criteria:

* Emergency surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Mean Near Infrared Saturation of the brain | Baseline within 5 minutes of intervention then Intraoperatively during intervention.
  Measure the NIRs of the brain by placeing NIRs monitoring patches on the forehead during clamped and unclamped intervention of the percutaneous superior vena cava line.

SECONDARY OUTCOMES:
Mean Blood Pressure | Intraoperatively during intervention.(every 5 minutes during 40 minute intervention period).
  Measure the Mean blood pressure during clamped/unclamped Percutaneous superior vena cava line placement.
Mean mixed venous saturation (non invasive measure) | Intraoperatively during intervention.(every 5 minutes during 40 minute intervention period).
  Measure the central venous ressure during clamped/unclamped intervention of percutaneous superior vena cava line.
CPB pump flow | Intraoperatively during intervention.(every 5 minutes during 40 minute intervention period).
  Measure the pump flow during clamped/unclamped intervention of percutaneous superior vena cava line.
Vacuum Pressure | Intraoperatively during intervention.(every 5 minutes during 40 minute intervention period).
  Measure the vacum pressure during clamped/unclamped intervention of percutaneous superior vena cava line.
Venous reservoir level | Intraoperatively during intervention.(every 5 minutes during 40 minute intervention period).
  Measure the venous reservoir level during clamped/unclamped intervention of percutaneous superior vena cava line.
Arterial blood gas | Initial, after first intervention arm(20 min), at end of study period (40 min)
  Measure arterial blood gases at baseline at after each intervention clamped(20 min)/unclamped (20 min) of percutaneous superior vena cava line.
Surgical visualization score | Baseline immediately before intervention period , end of each intervention period
  Score of 1-4 1=excellent visualization 4= poor visualization.
cerebral perfusion pressure | Intraoperatively during intervention.(every 5 minutes during 40 minute intervention period).
  Measure the cerebral perfusion pressure (MAP-CVP)during clamped/unclamped intervention of percutaneous superior vena cava line.
Central Venous Pressure | Intraoperatively during intervention.(every 5 minutes during 40 minute intervention period).
  Central venous pressure measured in the superior vena cava.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bainbridge, MD FRCPC, Principal Investigator — Lawson Health research institute, University of Western Ontario
Locations (1):
- London Health Sciences Centre, Univeristy Hospital, London, Ontario, Canada

REFERENCES:
- [Derived] Bainbridge DT, Chu MW, Kiaii B, Cleland A, Murkin J. Percutaneous superior vena cava drainage during minimally invasive mitral valve surgery: a randomized, crossover study. J Cardiothorac Vasc Anesth. 2015 Feb;29(1):101-6. doi: 10.1053/j.jvca.2014.07.020. Epub 2014 Nov 7. PMID 25440652